CLINICAL TRIAL: NCT05337033
Title: A Multi-Centre, Tolerability Study of a Cannabidiol-enriched Cannabis Herbal Extract for Chronic Headaches in Adolescents: the CAN-CHA Trial
Brief Title: Cannabis for Chronic Headaches in Adolescents: the CAN-CHA Trial
Acronym: CAN-CHA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: SickKids Foundation (Other)
Responsible Party: Principal Investigator, Lauren Kelly, Lauren E Kelly PhD, MSc, BMedSci, CCRP, Assistant Professor, Dept. of Pediatrics & Child Health, University of Manitoba Scientific Director, Canadian Childhood Cannabinoid Clinical Trials (www.C4Trials.org), University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN-CHA
Record Dates: First submitted 2022-03-29; First posted 2022-04-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Migraine
Keywords: Adolescents; Children; Cannabis; Migraine; Cannabidiol; Tetrahydrocannbinol
MeSH Terms: conditions — Marijuana Abuse; Migraine Disorders | interventions — Medical Marijuana

STUDY DESIGN:
Intervention Model Description: Open label tolerability trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cannabidiol-enriched Cannabis Herbal Extract (Experimental): CBD50 plus
  Interventions: Drug: MPL-001

INTERVENTIONS:
Drug: MPL-001 — CBD50 plus is a medical cannabis oil with flavouring agent produced under Good Manufacturing Practice by MediPharm Labs and purchased for this study. Each ml of oil contains 2 mg/ml of delta-9-THC and 50 mg/ml of CBD.
  Participants will receive escalating doses from 0.2-0.4 mg/kg/day of CBD to 0.8-1 mg/kg of CBD per day for four months, with dose increases monthly in 0.2mg/kg increments. Participants will following a weekly weaning protocol.
  Other Names: medical cannabis oil

SUMMARY:
Chronic headaches are a major cause of disability among adolescents. Cannabis products have supported the management of headaches in adults and may play a role in pediatric chronic pain. We propose a multisite, open-label, tolerability study conducted across three centers in Canada of Cannabidiol-enriched Cannabis Herbal Extract in adolescents (ages 14 to 17 years old) with chronic headaches. The study includes a one month baseline assessment, four months of escalating treatment doses and a weaning period. Our primary outcome is tolerability defined as the number and severity of reported adverse events.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Adolescents aged between 14-17 years of age at the time of screening.
2. Diagnosed with Chronic Migraine according to ICHD-3: headache (migraine-like or tension-type like) occurring on 15 or more days per month for more than 3 months which on at least 8 days per month have features of migraine headache. [121]
3. Failed at least two treatment options on the grounds of safety (tolerability) and/or efficacy, including but not limited to antidepressant (tricyclic antidepressant or selective norepinephrine reuptake inhibitor), magnesium, gabapentinoids topiramate and/or non-pharmacological therapies.
4. Females who have reached menarche should have a negative pregnancy test during screening.
5. Must be willing to engage with psychology and physiotherapy throughout the trial as appropriate.

Exclusion Criteria:

1. As per the investigator judgement, the participant is not an ideal candidate due to a personal issue or medical condition that is likely to impede in the successful completion of the study
2. Participants with a history of post-concussion headache or new daily persistent headache
3. Participants with a diagnosis of medication overuse headache
4. Participants with cardiac, renal or hepatic disease (assessed by the site investigator)
5. Participants with complex regional pain syndrome-II
6. Participants with abnormal ECG findings at baseline (as determined by the investigator)
7. Participants who are on the following medications: opioids, antipsychotics, antimanic, barbiturates, benzodiazepines, muscle relaxants, sedatives, or tramadol.
8. Participants with developmental delay or impairments including autism, cerebral palsy or intellectual disability.
9. Participants with a personal or family history of schizophrenia or psychotic disorders
10. Participants who are pregnant or breast/chest-feeding or plans to become pregnant within the study period or within three months of interventional product discontinuation
11. Participants who cannot commit to using contraception and refraining from recreational cannabis use and driving throughout the study period
12. Participants with known allergy to cannabinoids and/or palm/coconut oil

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cannabis-related adverse events | Reported daily through study completion, an average of 6 months
  The frequency of adverse events will be measured and characterized using standard CTCAE coding

SECONDARY OUTCOMES:
The frequency and duration of headache compared to baseline | Reported daily through study completion, an average of 6 months
  Reported headache frequency and duration daily and reported as a monthly average documented at baseline.
Pain intensity compared to baseline | Reported daily through study completion, an average of 6 months
  The average intensity measured using a Numeric Rating Scale (NRS) will be reported as a percentage change from the monthly average documented at baseline and an increasing score(highest score =10) indicates a greater severity of pain.
Pain impact on participants quality of life compared to baseline | Reported monthly for 6 months
  The impact of pain on participants quality of life using the PROMIS Pediatric Pain Interference- Short Form 8a will be reported as a percentage change from the monthly average documented at baseline.
Number of hours of sleep per night compared to baseline | Reported daily through study completion, an average of 6 months
  The number of hours of sleep per night will be measured using a actigraphy device
Change in sleep quality | Reported monthly for 6 months
  Patient Reported Outcome Measurement Information System (PROMIS) Pediatric Short Form v 2.0 - Pediatric Sleep-Related Impairment 8a scale as a percentage change from the monthly average documented at baseline where a higher number indicates a more sleep related impairment
Change in mood, depression from baseline | Reported monthly for 6 months
  PROMIS Pediatric Short Form v2.0 - Depressive Symptoms 8a scale as a percentage change from the monthly average documented at baseline
Change in mood, positive affect from baseline | Reported monthly for 6 months
  Change in mood, positive affect will be evaluated using PROMIS Pediatric Positive Affect - Short Form 8 and reported as a percentage change from the monthly average documented at baseline
Change in self-directed goal attainment from baseline | Reported monthly for 6 months
  Participants will self-directed goal attainment (participant and parent reported) as a percentage of goal attained at each study visit
Changes in anxiety compared to baseline | Reported monthly for 6 months
  Changes in anxiety will be measured using the PROMIS Pediatric Anxiety Short Form v2.0 and reported as percentage change from the monthly average documented at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Kelly, PhD, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University-, Halifax, Nova Scotia
  - North Toronto Neurology, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chhabra M, Lewis EC, Balshaw R, Stewart B, Zaslawski Z, Lowthian T, Alidina Z, Chesick-Gordis M, Xie W, Drogemoller BI, Wright GEB, Birnie KA, Boerner KE, Tsang VWL, Irwin SL, Pohl D, Weil AG, Sell E, Penz E, Robson-MacKay A, Mbabaali S, Blackman S, Gordon S, Alcorn J, Huntsman RJ, Oberlander TF, Finley GA, Kelly LE. A multi-centre, tolerability study of a cannabidiol-enriched Cannabis Herbal Extract for chronic headaches in adolescents: The CAN-CHA protocol. PLoS One. 2024 Sep 20;19(9):e0290185. doi: 10.1371/journal.pone.0290185. eCollection 2024. PMID 39302982